CLINICAL TRIAL: NCT07093372
Title: Comparison Between Laryngeal Mask and High-flow Nasal Oxygen Therapy in Obese Patients Undergoing Electroconvulsive Therapy
Brief Title: LMA vs High-flow Nasal Oxygen During ECT in Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eulji University Hospital (Other)
Responsible Party: Principal Investigator, Hyunjae Im, Assistant Professor of Anesthesiology and Pain Medicine, Eulji University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UEMC 2025-06-004-001
Record Dates: First submitted 2025-07-16; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Electroconvulsive Therapy Treated Patients; Obesity
Keywords: electroconvulsive therapy; obesity; ventilation strategy
MeSH Terms: conditions — Obesity | interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: All participants will undergo LMA in session 1 and 3, and HFNC in session 2 and 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alternating LMA and HFNC Oxygen Therapy (Experimental): All participants will undergo laryngeal mask airway (LMA) ventilation during ECT sessions 1 and 3, and high-flow nasal cannula (HFNC) oxygen therapy during sessions 2 and 4.
  Interventions: Device: Laryngeal Mask Airway; Device: High-Flow Nasal Cannula

INTERVENTIONS:
Device: Laryngeal Mask Airway — A supraglottic airway device (i-gel) used to deliver oxygen and assist ventilation during electroconvulsive therapy (ECT) in obese patients. The device is inserted after induction of general anesthesia and removed after spontaneous respiration is restored.
Device: High-Flow Nasal Cannula — A heated and humidified oxygen delivery system that provides high flow oxygen through nasal prongs. In this study, it is used throughout the ECT procedure to maintain oxygenation in obese patients without the need for invasive airway insertion.

SUMMARY:
This study aims to compare two oxygenation strategies-laryngeal mask airway (LMA) ventilation and high-flow nasal cannula (HFNC)-during electroconvulsive therapy (ECT) in obese patients. Due to their physiological characteristics, obese patients are at increased risk of hypoxia during ECT under general anesthesia.

Adult patients with a body mass index (BMI) ≥30 who are scheduled to undergo ECT will participate. Each participant will receive both oxygenation strategies in a fixed alternating order during four consecutive ECT sessions. The procedures will follow standard anesthesia protocols.

During the ECT procedures and the 30-minute recovery period in the post-anesthesia care unit, we will monitor the occurrence of hypoxia (SpO₂ <92%), ventilator parameters, vital signs, postoperative confusion within 24 hours, and any reports of dental discomfort. This information will help assess the safety and clinical utility of each oxygenation method for obese patients receiving ECT.

DETAILED DESCRIPTION:
Obesity is a known risk factor for perioperative hypoxia due to physiological changes such as increased airway resistance, reduced functional residual capacity, and elevated oxygen demand. These risks are amplified in patients undergoing electroconvulsive therapy (ECT) under general anesthesia, where periods of apnea can result in critical oxygen desaturation.

While laryngeal mask airways (LMAs) and high-flow nasal cannula (HFNC) therapy are both recommended strategies to maintain oxygenation during anesthesia, their comparative effectiveness in obese patients undergoing ECT has not been well established. LMAs provide direct airway access and enable positive pressure ventilation but carry a risk of dental trauma. HFNC offers a non-invasive alternative that may prolong safe apnea time, though its oxygenation efficacy during ECT remains unclear.

This study aims to evaluate the safety and effectiveness of LMA versus HFNC in preventing hypoxia during ECT in obese patients. Using a within-subject crossover design, each participant will receive both interventions in alternating ECT sessions. This trial will help determine the optimal airway management strategy for minimizing peri-procedural hypoxia in this high-risk population.

The outcome will be assessed during each ECT session as part of a crossover design. All participants will undergo both LMA and HFNC interventions in alternating sessions (LMA during sessions 1 and 3, HFNC during sessions 2 and 4). Oxygen support beyond the assigned method will be recorded when clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients scheduled to undergo ≥ 4 electroconvulsive therapy (ECT) sessions
* Body mass index (BMI) ≥ 30 kg/m² (WHO obesity classification)
* American Society of Anesthesiologists (ASA) physical status class I to III
* Provided written informed consent (by patient or legal guardian)

Exclusion Criteria:

* Patients under 18 years of age
* Patients with ASA class IV or V
* Patients with anticipated dental injury risk that precludes use of a laryngeal mask airway
* Patients or guardians who refuse participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia (SpO₂ <92%) during ECT | During each ECT session (approximately 10-15 minutes)

SECONDARY OUTCOMES:
incidence of hypoxia during recovery | During post-anesthesia recovery (approximately 30-40 minutes)
Lowest peripheral oxygen saturation | From preoxygenation to recovery room discharge (approximately 1 hours)
Duration of hypoxia during ECT and recovery | From preoxygenation to recovery room discharge (approximately 1 hours)
Lowest end-tidal CO₂ before ECT stimulation | Baseline (immediately prior to ECT stimulation)
Percent (%) increase in heart rate after ECT stimulation | During each ECT session (approximately 10-15 minutes)
Duration of seizure (motor and EEG) | During each ECT session (approximately 10-15 minutes)
Postictal Suppression Index (PSI) | During each ECT session (approximately 10-15 minutes)
Husain EEG Seizure Quality Scale | During each ECT session (approximately 10-15 minutes)
Airway management failure rate (LMA reinsertion or intubation required) | During each ECT session (approximately 10-15 minutes)
Number of participants with dental discomfort or tooth injury within 24 hours after ECT | Within 24 hours after each ECT session
Number of participants requiring additional oxygen support during ECT | During each ECT session (approximately 10-15 minutes)

IPD SHARING:
Plan to Share IPD: No